CLINICAL TRIAL: NCT06778499
Title: Effect of Plyometric Training on Lower Limbs Explosive Strength and Skill Performance Among University Student Latin Dancer in China
Brief Title: Effect of Plyometric Training on University Student Latin Dancers' Lower Limbs Explosive Strength and Skill Performance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, AI MENGQI, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AI MENGQI; 202501 (Registry Identifier: Protocol for plyometric training)
Record Dates: First submitted 2025-01-06; First posted 2025-01-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Physical Education and Training/Methods
Keywords: plyometric training; Explosive strength; Latin dancer; Latin dance performance
MeSH Terms: interventions — Plyometric Exercise; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training Protocol for Explosive Strength (Experimental): The experimental groups will undergo 3 interventions a week, with one session lasting 90 minutes. The experimental group will perform 15 minutes of dynamic stretching, 30 minutes of Latin dance-specific technique training, 30 minutes of plyometric training, and 15 minutes of relaxation stretching.
  Interventions: Other: Plyometric training for experimental group
- Traditional Training Protocol for Dance Performance (Experimental): The control group will perform 15 minutes of dynamic stretching, 30 minutes of Latin dance-specific technique training, 30 minutes of general training, and 15 minutes of relaxation stretching.
  Interventions: Other: Traditional training for control group

INTERVENTIONS:
Other: Plyometric training for experimental group — The experimental groups will undergo 3 interventions a week, with one session lasting 90 minutes. The experimental group will perform 15 minutes of dynamic stretching, 30 minutes of Latin dance-specific technique training, 30 minutes of plyometric training, and 15 minutes of relaxation stretching.
  Arms: Plyometric Training Protocol for Explosive Strength
Other: Traditional training for control group — The control group will perform 15 minutes of dynamic stretching, 30 minutes of Latin dance-specific technique training, 30 minutes of general training, and 15 minutes of relaxation stretching.
  Arms: Traditional Training Protocol for Dance Performance

SUMMARY:
The purpose of this study is to find out if plyometric training has an effect on lower limb explosive strength and skill performance in Latin dancers.

The aim is to answer the following questions:

1. Does augmented style training increase dancers' lower limb explosive strength.
2. Whether plyometric training promotes specialized dance skills.
3. The relationship between lower limb explosive strength and specialized dance skills.

The researchers set up an experimental group and a control group, the experimental group uses plyometric training and the control group performs traditional training, and finally, between-group and within-group comparisons are made.

Participants will:

Train for 90 minutes three times a week for eight weeks. Participants' lower limb explosive strength and skills will be measured before the start of the experiment and at the end of the experiment.

DETAILED DESCRIPTION:
1. Detailed Description The Intervention Protocol of this research used part of the research protocol of Chinese scholar Du Min (Du, 2020). This research utilized augmentative training as an intervention, with the dependent variables being the subject's lower limb explosive power and Latin dance skill performance. Through extensive literature review, countermovement jumps, standing long jump, and 20m-sprint were identified as measures of lower limb explosive power(Chen et al., 2023). The experimental and control groups will be tested on the same Cha Cha Dance Gold Medal solo routine and recorded with a video camera. Score athletic performance according to 'the Latin Dance Technical Quality Elements of the World DanceSport Federation（WDSF） 2.1 Evaluation System'. Lower limb explosive power is closely related to the skill performance of cha-cha dance, and the review of the relevant literature was determined to be posture, balance, footwork, preparation-movement-reduction, spinning and rotation, dynamic performance, and line extension as the test indicators of elementary skill (pei, 2023). In order to make the experiment more rigorous and scientific , to reduce the interference of uncontrollable factors , this research is Cluster Randomized Controlled Trial (CRCT) design , the students come from different areas . This experiment lasted for 8 weeks, 1.5 hours each time (Du, 2020), including one hour of physical fitness training and half an hour of specialized technical training. The sample was a population of university students who had been studying Latin dance for one year as well as more than one year, from Guangxi Normal University (Guilin) and Guilin University of Electronic Technology (Beihai), a total of 48 people. Dancers were randomly assigned to two different training locations and divided into experimental and control groups. Both groups will be trained in the Cha Cha Dance Single Gold Medal Moves. The experimental group will undergo plyometric training and the control group will undergo general training. This study measured the dependent variable three times throughout the intervention: baseline before the experimental intervention, post-test 1 after 4 weeks, and post-test 2 after 8 weeks. Finally, statistical analysis was conducted on the three test results.
2. Protocol Design The experiment will last a total of 8 weeks in order to familiarize the experimenter with the plyometric training protocol and to make the whole process more fluid. It is necessary to ensure correct technique during the jumping exercises to minimize the occurrence of injuries. This research will monitor heart rate to ensure that the training load is the same for the experimental group (plyometric training) and the control group (general training). Both groups will have the same heart rate for each session of training load from the preparation phase - training phase - stretching and relaxation phase during the intervention. The experimental and control groups will undergo 3 interventions a week, with one session lasting 90 minutes. The experimental group will perform 15 minutes of dynamic stretching, 30 minutes of Latin dance-specific technique training, 30 minutes of plyometric training, and 15 minutes of relaxation stretching. The control group will perform 15 minutes of dynamic stretching, 30 minutes of Latin dance-specific technique training, 30 minutes of general training, and 15 minutes of relaxation stretching.

ELIGIBILITY:
Inclusion Criteria:

1. Have at least one year and more hours of Latin dance study.
2. Must be a current university student.

Exclusion Criteria:

1. Athletes who were systematically training their explosive strength.
2. Athletes with sports injuries such as ankle or waist injuries who could not follow the entire training schedule for two months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Countermovement Jumps at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end.
  This parameter belongs to Explosive Strength. Participants test using either arm swing or crossed hips (without any arm swing) while performing vertical longitudinal jumps on a smart jumping mat. The participants in this research uses a cross-legged waist when performing both the pre-test and post-test. The Smart Jump Pad in this research has been performed to measure the performance of the CMJ by providing signals from the platform in an iPad 7,5 IOS 12.1.1). When the test equipment is ready, under the direction of the test administrator, the experimenter stands on the Smart Jump Mat and performs a vertical longitudinal jump. The experimenter jumps to the best of their ability and each jump was automatically recorded on the iPad. The unit is "cm". subjects will test three times and record the maximum height.
Change from baseline Standing Long Jumps at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end.
  This parameter belongs to Explosive Strength. Participants stand slightly apart in front of the jump line, bend their knees, and move their arms backwards, then swing their arms and jump as far as possible; Stand on both feet while maintaining an upright position. Measure the furthest horizontal distance. The unit is "cm". Participants will test two times and record the farthest distance.
Change from baseline 20m-sprint at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end.
  This parameter belongs to Explosive Strength. Use a stopwatch to record the duration of the participants' 30 m sprint. Set cones at 0 and 20 meters along a straight line. Participants place their toes on the starting line or behind the starting line, start from a stationary position, and sprint at maximum speed over the cone at a distance of 20 meters before safely slowing down. Test the time it takes to run a 20-meter sprint. The unit is "second(s)". Participants will test two times and record the fastest time from two tests.
Change from baseline Posture at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end.
  This parameter belongs to Dance Performance. Using a video camera, a recorded video of the Cha Cha Gold Medal solo routine is send to the 6 judges, and the pre- and post-tests need to be rated using the same criteria 'the Latin Dance Technical Quality Elements of World Dance Sport Federation (WDSF) 2.1 Evaluation System'.
  The score range is 1-10. These subjects are college students with a basic level of Latin dance, so a minimum score of 6 and a maximum score of 10 have been determined. There are three levels, very excellent (10 points), excellent (8 points), and average (6 points).
  The total score given by the six experts will be recorded and the average score will be calculated. The higher the score, the higher the level of Latin dance.
Change from baseline Balance at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end.
  This parameter belongs to Dance Performance. Using a video camera, a recorded video of the Cha Cha Gold Medal solo routine is send to the 6 judges, and the pre- and post-tests need to be rated using the same criteria 'the Latin Dance Technical Quality Elements of World Dance Sport Federation (WDSF) 2.1 Evaluation System'.
  The score range is 1-10. These subjects are college students with a basic level of Latin dance, so a minimum score of 6 and a maximum score of 10 have been determined. There are three levels, very excellent (10 points), excellent (8 points), and average (6 points).
  The total score given by the six experts will be recorded and the average score will be calculated. The higher the score, the higher the level of Latin dance.
Change from baseline Footwork at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end.
  This parameter belongs to Dance Performance. Using a video camera, a recorded video of the Cha Cha Gold Medal solo routine is send to the 6 judges, and the pre- and post-tests need to be rated using the same criteria 'the Latin Dance Technical Quality Elements of World Dance Sport Federation (WDSF) 2.1 Evaluation System'.
  The score range is 1-10. These subjects are college students with a basic level of Latin dance, so a minimum score of 6 and a maximum score of 10 have been determined. There are three levels, very excellent (10 points), excellent (8 points), and average (6 points).
  The total score given by the six experts will be recorded and the average score will be calculated. The higher the score, the higher the level of Latin dance.
Change from baseline Spins and Turns at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end.
  This parameter belongs to Dance Performance. Using a video camera, a recorded video of the Cha Cha Gold Medal solo routine is send to the 6 judges, and the pre- and post-tests need to be rated using the same criteria 'the Latin Dance Technical Quality Elements of World Dance Sport Federation (WDSF) 2.1 Evaluation System'.
  The score range is 1-10. These subjects are college students with a basic level of Latin dance, so a minimum score of 6 and a maximum score of 10 have been determined. There are three levels, very excellent (10 points), excellent (8 points), and average (6 points).
  The total score given by the six experts will be recorded and the average score will be calculated. The higher the score, the higher the level of Latin dance.
Change from baseline Preparation-movement-reduction at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end.
  This parameter belongs to Dance Performance. Using a video camera, a recorded video of the Cha Cha Gold Medal solo routine is send to the 6 judges, and the pre- and post-tests need to be rated using the same criteria 'the Latin Dance Technical Quality Elements of World Dance Sport Federation (WDSF) 2.1 Evaluation System'.
  The score range is 1-10. These subjects are college students with a basic level of Latin dance, so a minimum score of 6 and a maximum score of 10 have been determined. There are three levels, very excellent (10 points), excellent (8 points), and average (6 points).
  The total score given by the six experts will be recorded and the average score will be calculated. The higher the score, the higher the level of Latin dance.
Change from baseline Dynamic Performance at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end.
  This parameter belongs to Dance Performance. Using a video camera, a recorded video of the Cha Cha Gold Medal solo routine is send to the 6 judges, and the pre- and post-tests need to be rated using the same criteria 'the Latin Dance Technical Quality Elements of World Dance Sport Federation (WDSF) 2.1 Evaluation System'.
  The score range is 1-10. These subjects are college students with a basic level of Latin dance, so a minimum score of 6 and a maximum score of 10 have been determined. There are three levels, very excellent (10 points), excellent (8 points), and average (6 points).
  The total score given by the six experts will be recorded and the average score will be calculated. The higher the score, the higher the level of Latin dance.
Change from baseline Line Extension at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end.
  This parameter belongs to Dance Performance. Using a video camera, a recorded video of the Cha Cha Gold Medal solo routine is send to the 6 judges, and the pre- and post-tests need to be rated using the same criteria 'the Latin Dance Technical Quality Elements of World Dance Sport Federation (WDSF) 2.1 Evaluation System'.
  The score range is 1-10. These subjects are college students with a basic level of Latin dance, so a minimum score of 6 and a maximum score of 10 have been determined. There are three levels, very excellent (10 points), excellent (8 points), and average (6 points).
  The total score given by the six experts will be recorded and the average score will be calculated. The higher the score, the higher the level of Latin dance.

CONTACTS AND LOCATIONS:
Overall Officials: MENGQI AI, Principal Investigator — University Putra Malaysia

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I gradute

REFERENCES:
- [Background] Du, M. (2020). Effects of plyometric training on lower extremity explosive strength and athletic performance in adolescent Latin dancers (Master Dissertation). Beijing Sport University, Bei Jing.
- [Background] Effects of plyometric training on lower extremity explosive strength and athletic performance in adolescent Latin dancers
- See also: Academic websites in China — https://www.cnki.net/index/

DOCUMENTS (1):
  • Study Protocol (2025-01-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT06778499/Prot_000.pdf